CLINICAL TRIAL: NCT02215044
Title: A Phase I Open-label Dose-finding Study of Intravenous BI 2536 Administered in Repeated 4-week Cycles as Repeated Doses on Day 1 and Day 15 in Combination With Gemcitabine Administered on Day 1, Day 8 and Day 15 in Patients With Locally Advanced or Metastatic Pancreatic Cancer
Brief Title: Dose-finding Study of BI 2536 Administered in Combination With Gemcitabine in Patients With Locally Advanced or Metastatic Pancreatic Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1216.8
Record Dates: First submitted 2014-08-07; First posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — BI 2536; Gemcitabine

ARMS (1):
- BI 2536 in combination with gemcitabine (Experimental)
  Interventions: Drug: BI 2536, intravenous; Drug: Gemcitabine, intravenous

INTERVENTIONS:
Drug: BI 2536, intravenous
Drug: Gemcitabine, intravenous

SUMMARY:
Determination of the maximum tolerated dose (MTD), safety, and tolerability when BI 2536 was given on Day 1 and Day 15 in combination with gemcitabine given on Day 1, Day 8 and Day 15 every 28 days in patients with locally advanced or metastatic pancreatic adenocarcinoma and characterisation the antitumor activity, pharmacokinetic (PK) profile, and CA 19-9 tumor marker response in response to the combination of BI 2536 with gemcitabine in patients with locally advanced or metastatic pancreatic adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patient with histologically or cytologically confirmed locally advanced, unresectable or metastasized adenocarcinoma of the pancreas who:

  1. have not received gemcitabine chemotherapy for locally advanced or metastatic pancreatic cancer or
  2. have progressive disease not before at least 6 months from cessation of adjuvant gemcitabine chemotherapy following curative surgical tumor resection
* Male or female patient aged 18 years or older
* Life expectancy of at least three (3) months
* Eastern Co-operative Oncology Group (ECOG) performance score of 2 or less
* Patient must have given written informed consent

Exclusion Criteria:

* Prior chemo- (other than adjuvant gemcitabine), hormone- (other than Megace®) or immunotherapy
* Ampullary carcinoma of the pancreas
* Brain metastases, which are symptomatic or require therapy
* Patients who have any other life-threatening illness or organ system dysfunction, which in the opinion of the investigator, would either compromise patient safety or interfere with the evaluation of the safety of the test drug
* Other malignancies diagnosed within the past five (5) years (other than non-melanomatous skin cancer)
* Absolute neutrophil count (ANC) <1,500/μl, platelet count <150,000/μl, or hemoglobin <9 g/dl
* Total bilirubin >1.8mg/dl (>30.78 μmol/l,, international system of units (SI) equivalent) under adequate drainage measures (in case of obstructive jaundice)
* No hepatic metastases: Aspartate amino transferase (AST) and/or alanine amino transferase (ALT) >2.5 x upper limit of normal (ULN). Hepatic metastases: aspartate amino transferase (AST) and/or alanine amino transferase (ALT) >5 x ULN
* Serum creatinine >2.0 mg/dl (>176 μmol/L, SI Unit equivalent)
* Radiotherapy within the last 2 weeks prior to or during treatment with the trial drug
* Patients with any serious active infection (i.e., requiring an IV antibiotic, antifungal, or antiviral agents)
* Patients with known HIV, Hepatitis-B or -C infection
* Known or suspected active drug or alcohol abuse
* Women of child-bearing potential; men who are able to father a child and are unwilling to use a medically acceptable method of contraception during the trial
* Pregnancy or breast feeding
* Treatment with any investigational drug within the past 4 weeks or within less than four half-life times of the investigational drug before treatment with the trial drug and/or persistence of toxicities of prior anticancer therapies which are deemed to be clinically relevant
* Patient unable to comply with the protocol
* Patients requiring warfarin (Coumadin®) or patients with a known pre-existing coagulopathy unrelated to pancreatic cancer (This means, for example, that patient with a long (years) history or recurrent venocclusive disease clearly preceding the diagnosis of pancreatic cancer will be excluded from the study. Patients with recent hypercoagulable state (ie deep vein thrombosis or pulmonary embolism) due to pancreatic cancer who are clinically stable on low molecular weight heparin will not be excluded)
* Patients with neuropathy (sensory or motor) ≥ common terminology criteria for adverse events (CTCAE) 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-06; Primary Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Occurence of dose limiting toxicity according to CTCAE | up to day 28 of each cycle

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analytes in plasma from time zero to infinity (AUC0-∞) | Pre-dose, up to 192 hours after start of treatment
Maximum measured concentration of the analytes in plasma (Cmax) | Pre-dose, up to 192 hours after start of treatment
Objective tumour responses based on Response evaluation criteria in solid tumors (RECIST) criteria | up to 1 year
Survival status | up to 1 year
Tumor marker (CA19-9) response to treatment with BI 2536 and gemcitabine | Day 1 of each treatment cycle prior to administration of study treatment